CLINICAL TRIAL: NCT01157234
Title: Nebivolol Effect on Nitric Oxide Levels, Blood Pressure, and Renal Function in Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BYS-MD-42
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
Keywords: Hypertension; Kidney transplantation; Renal function; Nitric Oxide; Nebivolol
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Active Comparator): Nebivolol starting dose of 5 mg orally once daily, titrated to a maximum total daily dose of 40 mg daily to achieve a target blood pressure of <140/90 and continued until month-12 of the study.
  Interventions: Drug: Nebivolol
- Metoprolol (Active Comparator): Metoprolol starting dose of 25mg orally once twice daily, titrated to a maximum total daily dose of 400 mg to achieve a target blood pressure of <140/90 and continued until month-12 of the study.
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 5 mg once daily, titrated to a maximum total daily dose of 40 mg to achieve a blood pressure of < 140/ 90.
  Other Names: Bystolic
  Arms: Nebivolol
Drug: Metoprolol — Metoprolol 25 mg twice daily, titrated to a maximum total daily dose of 400 mg to achieve a blood pressure < 140/90.
  Other Names: Lopressor
  Arms: Metoprolol

SUMMARY:
This study will investigate the blood pressure lowering efficacy of nebivolol among renal transplant recipients who are on calcineurin inhibitors which are believed to contribute to hypertension by sympathetic nervous system (SNS) activation and decreased prostaglandin and nitric oxide production. Hypotheses:

1. There is a significant difference in the effect of 12 months of Nebivolol versus Metoprolol treatment on the plasma nitric oxide level of hypertensive renal transplant patients.
2. There is a significant difference in the effect of 12 months of Nebivolol versus Metoprolol treatment on the estimated glomerular filtration rate of hypertensive renal transplant patients.
3. There is a significant difference in the effect of 12 months of Nebivolol versus Metoprolol treatment on the systolic, diastolic and mean arterial blood pressures of hypertensive renal transplant patients.

DETAILED DESCRIPTION:
Nitric Oxide (NO) plays a plethora of functions in the kidney including vascular and hemodynamic regulation, fluid and electrolyte transport, and is an important component of pressure natriuresis and tubule-glomerular feedback.

Deficient NO levels have been associated with oxidative stress in conditions like hypertension, diabetes mellitus, and cardiovascular disease. NO deficiency has been identified in states of chronic progressive renal disease and altered NO production and/or decreased bioavailability is believed to characterize the endothelial dysfunction and resistant hypertension of renal failure.

It has been shown that kidney transplantation improves endothelium-dependent vasodilation in patients with end-stage renal disease (ESRD) and the NO activity significantly increases after transplantation. However, calcineurin inhibitor drugs used in the anti-rejection regimen can reduce endothelial NO production and aggravate hypertension through vascular and renal mechanisms. In turn, uncontrolled elevation in blood pressure has been associated with increased renal allograft failure and post-transplant mortality.

In the absence of randomized clinical trials of antihypertensive drugs and optimal blood pressure goals in kidney transplant recipients. There is no scientifically-robust consensus on the specific drugs to use among transplant patients. Nebivolol, is a third generation B1-selective B-blocker shown to have similar BP-lowering effect as other B-blockers, angiotensin converting enzyme (ACE) inhibitors and angiotensin II receptor blocker (ARB) drugs, and calcium channel blockers. Nebivolol ameliorates hypertension by increasing NO release, promoting arterial and venous vasodilatation and beta-blockade. Nebivolol has beneficial effect on the kidney allograft. Studies in animal transplants have shown that nebivolol could reduce ischemia-induced reperfusion injury, alleviate renal perfusion pressure and increase NO release with associated vasodilation of the renal vasculature. These effects have not been seen with older generation B-blockers like propranolol or bisoprolol. Finally, in surgically reduced renal mass, nebivolol has been demonstrated to attenuate collagen type 1 expression with lessening of glomerular and interstitial fibrosis.

In this study, the effect of nebivolol and metoprolol on the change in NO level at baseline and at the 12th month of treatment will be compared. Similarly,the effects of the two drugs on the change in renal function, blood pressure, and blood pressure regimen from baseline to month-12 of treatment will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age who are recipients of - a solitary kidney or combined kidney-pancreas transplant within the last twenty four months
* Current diagnosis of hypertension
* Normal hepatic enzymes
* Estimated creatinine clearance (by cockcroft-gault formula) >or= 30 ml/min

Exclusion Criteria:

* Any contraindication to taking beta-blockers, specifically Nebivolol or Metoprolol. Conditions such as : (bradycardia heart rate (HR) <60 beats per minute , heart block > 1st degree, decompensated cardiac failure, sick sinus syndrome (unless permanent pacemaker in place), severe hepatic impairment( defined as elevation of aspartamine aminotransferase , alanine aminotransferase, or bilirubin levels to three times upper limit of normal reference range), severe peripheral arterial circulatory disorder, history of bronchospasm and /or asthma and /or regular medication with inhaled bronchodilators. or , or any medical condition that in the opinion of the investigator may interfere with the subject's ability to successfully complete the protocol.
* Any medical condition which, in the opinion of the Principal Investigator, might compromise the safety of the subject in participating in the protocol such as hypotension or not requiring antihypertensive medications.
* Any serious systemic disease that might complicate management and reduce life expectancy.
* Uncontrolled hypertension defined as systolic blood pressure (SBP) > 210 or diastolic blood pressure (DBP) > 120 mm Hg.
* Symptomatic hypotension
* Previous intolerance to beta blockers
* Cerebrovascular accident within 3 months of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Santos, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Schmidt RJ, Yokota S, Tracy TS, Sorkin MI, Baylis C. Nitric oxide production is low in end-stage renal disease patients on peritoneal dialysis. Am J Physiol. 1999 May;276(5):F794-7. doi: 10.1152/ajprenal.1999.276.5.F794. PMID 10330062
- [Background] Uzun H, Konukoglu D, Besler M, Erdenen F, Sezgin C, Muderrisoglu C. The effects of renal replacement therapy on plasma, asymmetric dimethylarginine, nitric oxide and C-reactive protein levels. Clin Invest Med. 2008;31(1):E1-7. doi: 10.25011/cim.v31i1.3135. PMID 18312743
- [Background] Passauer J, Bussemaker E, Lassig G, Gross P. Kidney transplantation improves endothelium-dependent vasodilation in patients with endstage renal disease. Transplantation. 2003 Jun 15;75(11):1907-10. doi: 10.1097/01.TP.0000065739.19681.93. PMID 12811255
- [Background] Zhang W, Zhou C, Xie J, Chen B, Chang L. Serum asymmetric dimethylarginine and endothelial function after renal transplantation. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2009 Apr;34(4):289-94. PMID 19411743
- [Background] Schwenger V, Zeier M, Ritz E. Hypertension after renal transplantation. Ann Transplant. 2001;6(4):25-30. PMID 12035455
- [Background] Opelz G, Wujciak T, Ritz E. Association of chronic kidney graft failure with recipient blood pressure. Collaborative Transplant Study. Kidney Int. 1998 Jan;53(1):217-22. doi: 10.1046/j.1523-1755.1998.00744.x. PMID 9453022
- [Background] Curtis JJ, Luke RG, Jones P, Diethelm AG. Hypertension in cyclosporine-treated renal transplant recipients is sodium dependent. Am J Med. 1988 Aug;85(2):134-8. doi: 10.1016/s0002-9343(88)80331-0. PMID 3041828
- [Background] Koomans HA, Ligtenberg G. Mechanisms and consequences of arterial hypertension after renal transplantation. Transplantation. 2001 Sep 27;72(6 Suppl):S9-12. doi: 10.1097/00007890-200109271-00004. PMID 11585243
- [Background] Ojo AO. Cardiovascular complications after renal transplantation and their prevention. Transplantation. 2006 Sep 15;82(5):603-11. doi: 10.1097/01.tp.0000235527.81917.fe. PMID 16969281
- [Background] Cheng JW. Nebivolol: a third-generation beta-blocker for hypertension. Clin Ther. 2009 Mar;31(3):447-62. doi: 10.1016/j.clinthera.2009.03.007. PMID 19393838
- [Background] Ignarro LJ. Experimental evidences of nitric oxide-dependent vasodilatory activity of nebivolol, a third-generation beta-blocker. Blood Press Suppl. 2004 Oct;1:2-16. PMID 15587107
- [Background] Kamp O, Sieswerda GT, Visser CA. Comparison of effects on systolic and diastolic left ventricular function of nebivolol versus atenolol in patients with uncomplicated essential hypertension. Am J Cardiol. 2003 Aug 1;92(3):344-8. doi: 10.1016/s0002-9149(03)00645-3. PMID 12888152
- [Background] Brehm BR, Wolf SC, Bertsch D, Klaussner M, Wesselborg S, Schuler S, Schulze-Osthoff K. Effects of nebivolol on proliferation and apoptosis of human coronary artery smooth muscle and endothelial cells. Cardiovasc Res. 2001 Feb 1;49(2):430-9. doi: 10.1016/s0008-6363(00)00253-4. PMID 11164853
- [Background] Gandhi C, Zalawadia R, Balaraman R. Nebivolol reduces experimentally induced warm renal ischemia reperfusion injury in rats. Ren Fail. 2008;30(9):921-30. doi: 10.1080/08860220802353900. PMID 18925533
- [Background] Georgescu A, Pluteanu F, Flonta ML, Badila E, Dorobantu M, Popov D. The cellular mechanisms involved in the vasodilator effect of nebivolol on the renal artery. Eur J Pharmacol. 2005 Jan 31;508(1-3):159-66. doi: 10.1016/j.ejphar.2004.11.043. Epub 2005 Jan 7. PMID 15680267
- [Background] Kakoki M, Hirata Y, Hayakawa H, Nishimatsu H, Suzuki Y, Nagata D, Suzuki E, Kikuchi K, Nagano T, Omata M. Effects of vasodilatory beta-adrenoceptor antagonists on endothelium-derived nitric oxide release in rat kidney. Hypertension. 1999 Jan;33(1 Pt 2):467-71. doi: 10.1161/01.hyp.33.1.467. PMID 9931149
- [Background] Pires MJ, Rodriguez-Pena AB, Arevalo M, Cenador B, Evangelista S, Esteller A, Sanchez-Rodriguez A, Colaco A, Lopez-Novoa JM. Long-term nebivolol administration reduces renal fibrosis and prevents endothelial dysfunction in rats with hypertension induced by renal mass reduction. J Hypertens. 2007 Dec;25(12):2486-96. doi: 10.1097/HJH.0b013e3282efeecb. PMID 17984671
- [Background] Meier-Kriesche HU, Schold JD, Kaplan B. Long-term renal allograft survival: have we made significant progress or is it time to rethink our analytic and therapeutic strategies? Am J Transplant. 2004 Aug;4(8):1289-95. doi: 10.1111/j.1600-6143.2004.00515.x. PMID 15268730
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at the University of Florida and Shands Renal Transplant Clinic.
  The first patient was randomized on July 8, 2010 and the follow up of the last patient ended on July 21, 2014.
Pre-assignment Details: 32 participants were screened, 2 failed screening and 30 met the eligibility criteria and randomized to either the arm with nebivolol or the arm with metoprolol.
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who signed informed consent and received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (15.9) | 46.4 (13.8) | 49.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Plasma Nitric Oxide [Mean (Standard Deviation); unit: nmol/l] — Full analysis included all participants who signed informed consent and received at least one dose of study drug.
  nmol/l | 52.93 (21.09) | 48.23 (15.37) | 50.53 (17.99)
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: milliliter/minute] — Estimated glomerular filtration rate is calculated according to the modification of diet in renal disease equation using age, gender and race in calculating kidney function.
  Full analysis included all participants who signed informed consent and received at least one dose of study drug
  milliliter/minute | 53.13 (14.15) | 54.47 (14.65) | 53.80 (13.67)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeter, mercury] — Full analysis included all participants who signed informed consent and received at least one dose of study drug.
  millimeter, mercury | 132.93 (15.79) | 131.33 (18.14) | 132.13 (16.73)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeter, mercury] — Full analysis included all participants who signed informed consent and received at least one dose of study drug
  millimeter, mercury | 84.07 (8.59) | 86.33 (8.62) | 85.20 (8.53)
Mean Arterial Blood Pressure [Mean (Standard Deviation); unit: millimeter, mercury] — Full analysis included all participants who signed informed consent and received at least one dose of study drug
  millimeter, mercury | 100.20 (8.06) | 101.47 (10.76) | 100.83 (9.36)
Number of Antihypertensive Drug Classes Being Used [Mean (Standard Deviation); unit: Antihypertensive Drug Classes] — Full analysis included all participants who signed informed consent and received at least one dose of study drug
  Antihypertensive Drug Classes | 2.00 (0.84) | 1.80 (0.68) | 1.90 (0.89)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Nitric Oxide Level Change From Baseline to Month 12 Between the Groups.
Description: Percent change in Nitric Oxide (NO) blood level (nmol/L)=[Month-12 NO blood level minus baseline NO blood level] divided by [baseline NO blood level] multiplied by 100, where all levels are in nmol/L.
Time Frame: Change in Baseline, Month-12
Population: Full analysis set included all participants who signed informed consent and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 15 | 15
percent change | 11.47 (9.20) | -17.27 (9.20)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol; Test type: Superiority or Other; Least Squares Mean Difference = 28.73, 95.00% CI 2-sided [1.93 to 55.53]

2. Secondary Outcome: Estimated Glomerular Filtration Rate (ml/Minute) Change From Baseline to Month-12 Between the Groups
Description: The changed percentage in Estimated Glomerular Filtration Rate (eGFR), (based on the Modification of Diet in Renal Disease Equation)=[Month-12 GFR level minus baseline eGFR level] divided by [baseline eGFR level] multiplied by 100, where all levels are in ml/min.
Time Frame: Change in Baseline, Month-12
Population: Full analysis set included all participants who signed inform consent and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 15 | 15
percent change | 2.16 (7.16) | 10.43 (7.16)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol; Test type: Superiority or Other; Least Squares Mean Difference = 8.27, 95% CI 2-sided [-12.58 to 29.12]

3. Secondary Outcome: Systolic Blood Pressure (Millimeter, Mercury) Change From Baseline to Month-12 of Treatment Between the Groups
Description: Absolute change in Systolic Blood Pressure (SBP), (millimeter, Mercury)=Month-12 sitting trough SBP level minus baseline sitting trough SBP level
Time Frame: Change in Baseline, Month-12
Population: Full analysis set included all participants who signed inform consent and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: millimeter, Mercury
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 15 | 15
millimeter, Mercury | -2.65 (2.73) | -3.88 (2.73)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol; Test type: Superiority or Other; Least squares mean difference = 1.23, 95% CI 2-sided [-6.74 to 9.20], Standard Error of Mean 3.87

4. Secondary Outcome: Diastolic Blood Pressure (Millimeter, Mercury) Change From Baseline to Month-12 Between the Groups
Description: Absolute Change in Diastolic Blood Pressure (DBP), (millimeter, Mercury)= Month-12 sitting trough Diastolic Blood Pressure (millimeter, Mercury) level minus baseline sitting trough Diastolic Blood Pressure (millimeter, Mercury).
Time Frame: Change in Baseline, Month-12
Population: Full analysis set included all participants who signed inform consent and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: millimeter, mercury
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 15 | 15
millimeter, mercury | -0.66 (1.91) | -2.35 (1.91)

5. Secondary Outcome: Mean Arterial Blood Pressure (Millimeter, Mercury) Change From Baseline to Month-12 Between the Groups
Description: Absolute change in Mean Arterial Blood Pressure, (MAP), (millimeter, Mercury= Month-12 sitting trough MAP minus baseline sitting trough MAP.
  Mean Arterial Pressure= 2/3 trough diastolic blood pressure + 1/3 trough systolic blood pressure
Time Frame: Change in Baseline, Month-12
Population: Full analysis set included all participants who signed inform consent and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: millimeter, Mercury
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 15 | 15
millimeter, Mercury | -1.07 (2.11) | -3.19 (2.11)

6. Secondary Outcome: Number of Antihypertensive Drug Classes Change From Baseline to Month-12 Between the Groups.
Description: Percent change in quantity of Anti-Hypertensive Drug Classes (AHDC)=[Month-12 absolute number of AHDC minus baseline absolute number of AHDC] divided by [baseline absolute number of AHDC] multiplied by 100.
Time Frame: Change in Baseline, Month-12
Population: Percent change
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 15 | 15
percent change | -8.14 (11.58) | 8.70 (11.58)

7. Other Pre Specified Outcome: Plasma Nitric Oxide Level (Nmol/L) at Month-12 Between the Groups.
Time Frame: 12 Months
Population: Full analysis set included all participants who signed inform consent and received at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 15 | 15
nmol/L | 50.07 (3.93) | 38.13 (3.93)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol; Test type: Superiority or Other; Least Squares Mean Difference = 11.94, 95.00% CI 2-sided [0.48 to 23.40]

8. Post Hoc Outcome: Percent Change in Plasma Nitric Oxide Level From Baseline to Month-12 of Treatment With Nebivolol in Transplant Recipients <50 Years Old Compared With Metoprolol in Transplant Recipients >/= 50 Years Old.
Time Frame: Baseline and Month-12
Population: Nebivolol and metoprolol groups were subdivided into <50 years old and >50 years old subgroups and differences between subgroups were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Nebivolol <50 Year Old: Hypertensive kidney transplant recipients less than 50 years of age treated with Nebivolol starting dose of 5 mg orally once daily, titrated to a maximum total daily dose of 40 mg daily to achieve a target blood pressure of <140/90 and continued until month-12 of the study
- Metoprolol >/= 50 Year Old: Hypertensive kidney transplant recipients age 50 years or higher treated with Metoprolol starting dose of 5 mg orally once daily, titrated to a maximum total daily dose of 40 mg daily to achieve a target blood pressure of <140/90 and continued until month-12 of the study
Arm/Group | Nebivolol <50 Year Old | Metoprolol >/= 50 Year Old
Number analyzed (Participants) | 6 | 7
percent change | 51.55 (14.55) | -17.99 (13.47)
Statistical Analysis 1: Comparison: Nebivolol <50 Year Old vs Metoprolol >/= 50 Year Old; Test type: Superiority or Other; Least Squares Mean Difference = 69.54, 99.7% CI 2-sided [12.71 to 126.37], Standard Error of Mean 19.83

9. Post Hoc Outcome: Percent Change in Plasma Nitric Oxide Level From Baseline to Month-12 of Treatment With Nebivolol in Transplant Recipients < 50 Years Old Compared With Metoprolol in Transplant Recipients < 50 Years Old
Time Frame: Change in Baseline, Month-12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Nebivolol < 50 Years Old: Hypertensive kidney transplant recipients less than 50 years of age treated with Nebivolol starting dose of 5 mg orally once daily, titrated to a maximum total daily dose of 40 mg daily to achieve a target blood pressure of <140/90 and continued until month-12 of the study.
- Metoprolol <50 Years Old: Hypertensive kidney transplant recipients less than 50 years of age treated with Metoprolol starting dose of 25mg orally once twice daily, titrated to a maximum total daily dose of 400 mg to achieve a target blood pressure of <140/90 and continued until month-12 of the study.
Arm/Group | Nebivolol < 50 Years Old | Metoprolol <50 Years Old
Number analyzed (Participants) | 6 | 8
percent change | 51.55 (14.55) | -16.64 (12.60)
Statistical Analysis 1: Comparison: Nebivolol < 50 Years Old vs Metoprolol <50 Years Old; Test type: Superiority or Other; Least Squares Mean Difference = 68.19, 99.17% CI 2-sided [13.02 to 123.36], Standard Error of Mean 19.24

10. Post Hoc Outcome: Percent Change in Plasma Nitric Oxide Level From Baseline to Month-twelve of Treatment With Nebivolol in Transplant Recipients >/= 50 Years Old Compared With Nebivolol in Transplant Recipients < 50 Years Old.
Time Frame: Change in Baseline, Month-12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Nebivolol >/=50 Years Old: Hypertensive kidney transplant recipients age 50 years or higher treated with Nebivolol starting dose of 5 mg orally once daily, titrated to a maximum total daily dose of 40 mg daily to achieve a target blood pressure of <140/90 and continued until month-12 of the study.
- Metoprolol <50 Years Old: Hypertensive kidney transplant recipients age less than 50 years treated with Metoprolol starting dose of 25mg orally once twice daily, titrated to a maximum total daily dose of 400 mg to achieve a target blood pressure of <140/90 and continued until month-12 of the study.
Arm/Group | Nebivolol >/=50 Years Old | Metoprolol <50 Years Old
Number analyzed (Participants) | 9 | 8
percent change | -15.25 (11.88) | -16.64 (12.60)
Statistical Analysis 1: Comparison: Nebivolol >/=50 Years Old vs Metoprolol <50 Years Old; Test type: Superiority or Other; Least Squares Mean Difference = 1.39, 99.17% CI 2-sided [-48.25 to 51.03], Standard Error of Mean 17.32

11. Post Hoc Outcome: Percent Change in Plasma Nitric Oxide Level From Baseline to Month-12 of Treatment With Nebivolol in Transplant Recipients >/= 50 Years Old Compared With Metoprolol in Transplant Recipients Age >/= 50 Years Old.
Time Frame: Change in Baseline, Month-12
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Metoprolol >/=50 Years Old: Hypertensive kidney transplant recipients age 50 years or higher treated with Metoprolol starting dose of 25mg orally once twice daily, titrated to a maximum total daily dose of 400 mg to achieve a target blood pressure of <140/90 and continued until month-12 of the study.
Arm/Group | Nebivolol >/=50 Years Old | Metoprolol >/=50 Years Old
Number analyzed (Participants) | 9 | 7
percent change | -15.25 (11.88) | -17.99 (13.47)
Statistical Analysis 1: Comparison: Nebivolol >/=50 Years Old vs Metoprolol >/=50 Years Old; Test type: Superiority or Other; Least Squares Mean Difference = 2.74, 99.17% CI 2-sided [-48.74 to 54.22], Standard Error of Mean 17.96

12. Secondary Outcome: Plasma Asymmetric Dimethylarginine (ADMA) Change From Baseline to Month 12 Between the Groups
Description: Percent change in plasma ADMA (umol/L)=[month-12 plasma ADMA level minus baseline plasma ADMA level] divided by [baseline plasma ADMA level] multiplied by 100, where all levels are in umol/L.
Time Frame: Baseline, Month-12
Population: Technical limitations constrained measurements of Asymmetric Dimethylarginine (ADMA), resulting in no analysis for this outcome.
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Plasma Arginine (ARG) Level Change From Baseline to Month-12 Between Groups
Description: Percent change in plasma Arginine (umol/L)=[month-12 plasma Arginine level minus baseline plasma Arginine level] divided by [baseline plasma Arginine level] multiplied by 100, where all levels are in umol/L
Time Frame: Baseline, Month-12
Population: Technical limitations constrained measurements of plasma Arginine, resulting in no analysis for this outcome.
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Nebivolol | Metoprolol
Serious Adverse Events (participants affected / at risk) | 4/15 | 5/15
Other Adverse Events (participants affected / at risk) | 9/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=15) | Metoprolol (N=15)
Urinary Tract Infection (Infections and infestations) | 1 | 0
Abdominal Hematoma (Injury, poisoning and procedural complications) | 1 | 0
Renal Insufficiency (Renal and urinary disorders) | 2 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Herniorraphy (Surgical and medical procedures) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cytomegalovirus Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=15) | Metoprolol (N=15)
leukopenia (Blood and lymphatic system disorders) | 0 | 1
hyperglycemia (Endocrine disorders) | 2 | 3
Earache (Ear and labyrinth disorders) | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Chest Pain (General disorders) | 1 | 1
Edema (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Influenza-like Illness (General disorders) | 1 | 0
Cytomegalovirus Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 3
Arm Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Hydrocele (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed in a single center limits precision and generalizability of results.

Technical limitations prevented measurements of asymmetric dimethyl-arginine and arginine leading to absence of analysis for these outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other